CLINICAL TRIAL: NCT01444001
Title: Study of an Investigational Pneumococcal Vaccine in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PPR01
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-09

CONDITIONS: Pneumococcal Infections; Pneumococcal Pneumonia
Keywords: Pneumococcal Infections; Pneumococcal Vaccines; pneumococcal protein
MeSH Terms: conditions — Pneumococcal Infections; Pneumonia, Pneumococcal | interventions — Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pneumococcal Vaccine Dose 1 (Low dose) (Experimental): Participants will receive 2 injections of Dose 1 investigational Pneumococcal vaccine (Low dose) on Day 0 and Day 30, respectively.
  Interventions: Biological: Pneumococcal Vaccine
- Pneumococcal Vaccine Dose 2 (Middle dose) (Experimental): Participants will receive 2 injections of the investigational Pneumococcal vaccine (Middle dose) on Day 0 and Day 30, respectively.
  Interventions: Biological: Pneumococcal Vaccine
- Pneumococcal Vaccine Dose 3 (High dose) (Experimental): Participants will receive 2 injections of the investigational Pneumococcal vaccine (High dose) on Day 0 and Day 30, respectively.
  Interventions: Biological: Pneumococcal Vaccine

INTERVENTIONS:
Biological: Pneumococcal Vaccine — 0.5 mL, intramuscular
  Arms: Pneumococcal Vaccine Dose 1 (Low dose)
Biological: Pneumococcal Vaccine — 0.5 mL, intramuscular
  Arms: Pneumococcal Vaccine Dose 2 (Middle dose)
Biological: Pneumococcal Vaccine — 0.5 mL, intramuscular
  Arms: Pneumococcal Vaccine Dose 3 (High dose)

SUMMARY:
This study was designed to evaluate the safety, tolerability, and immunogenicity of three doses of an investigational pneumococcal vaccine in healthy adult volunteers.

Primary Objective:

* To evaluate the safety and tolerability of an investigational Pneumococcal vaccine.

DETAILED DESCRIPTION:
Each volunteer participant will receive two injections with one of three vaccine doses, administered on Day 0 and Day 30, in a dose-ascending manner, pending safety review at each dose level. All participants will be monitored for safety for 30 days after each injection.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 50 years on the day of inclusion
* Healthy, as determined by medical history and clinical examination
* Informed consent obtained
* Able to attend all scheduled visits and to comply with all trial procedures
* For a woman, inability to bear a child or negative urine pregnancy test at each vaccination visit
* For a woman of child-bearing potential: use of two medically acceptable, effective methods of contraception (oral contraceptive, intrauterine device, diaphragm, spermicide, or condom) or abstinence throughout the study participation starting at least 30 days prior to the first vaccination up to at least 30 days after the last vaccination.

Exclusion Criteria:

* Serious chronic disease (i.e., cardiac, renal, neurologic, rheumatologic, metabolic, gastrointestinal, psychiatric, or other organ system) that could interfere with trial conduct or and/or raise a safety concern
* For a woman, breast-feeding
* Participation in another clinical trial in the 30 days preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy
* Systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances
* Current abuse of alcohol or drug addiction that may interfere with the subject's ability to comply with trial procedures
* Blood or blood-derived products received in the past 3 months
* Any vaccination in the 30 days preceding the first trial vaccination
* Vaccination planned in the 30 days following any trial vaccination
* Known Human Immunodeficiency Virus (HIV), hepatitis B, or hepatitis C seropositivity
* Known thrombocytopenia or bleeding disorder contraindicating intramuscular (IM) vaccination
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent
* Febrile illness (≥ 38.0°C [or 100.4°F]) within 72 hours of inclusion/vaccination
* Previous vaccination in the preceding 5 years against pneumococcal disease with another vaccine
* History of pneumococcal infection (confirmed either clinically, serologically, or microbiologically) within 5 years
* Subject at high risk of pneumococcal infection during the trial
* Subjects living in a household with children < 5 years of age
* Antibiotic usage or upper or lower respiratory tract infection within one week before any blood draw for immunogenicity (Visits 1, 3, and 5).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2007-02; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The occurrence of solicited injection site reactions, solicited systemic reactions, unsolicited systemic reactions, and serious adverse events occurring throughout the trial | Day 0 up to Day 60 post vaccination
  Solicited injection site reactions: Pain, Erythema, and Swelling. Solicited systemic reactions: Fever (Temperature), Headache, Malaise, and Myalgia

SECONDARY OUTCOMES:
Immunogenicity of pneumococcal vaccine after 2 vaccinations | Day 0 and 30 days post vaccination
  Evaluation of immune responses to antigen component of the investigational vaccine by enzyme linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Ltd.
Locations (1):
- Allschwil, Switzerland

REFERENCES:
- [Derived] Seiberling M, Bologa M, Brookes R, Ochs M, Go K, Neveu D, Kamtchoua T, Lashley P, Yuan T, Gurunathan S. Safety and immunogenicity of a pneumococcal histidine triad protein D vaccine candidate in adults. Vaccine. 2012 Dec 14;30(52):7455-60. doi: 10.1016/j.vaccine.2012.10.080. Epub 2012 Nov 3. PMID 23131206
- See also: Related Info — http://www.sanofipasteur.com